CLINICAL TRIAL: NCT04960410
Title: Real Time Early Warning Model and Mobile Medical Assistant System for the Impact of Air Pollution on Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Real Time Early Warning Model and Mobile Medical Assistant System for the Impact of Air Pollution on AECOPD Disease
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beihang University (Other)
Responsible Party: Sponsor
Other Study IDs: LM2018072
Record Dates: First submitted 2021-07-04; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low air pollution
  Interventions: Combination Product: Types and exposure of different air pollutants
- High air pollution
  Interventions: Combination Product: Types and exposure of different air pollutants

INTERVENTIONS:
Combination Product: Types and exposure of different air pollutants — Types and exposure of different air pollutants in COPD patients' living and working environment

SUMMARY:
Objective to establish a real-time early warning model of acute exacerbation of chronic obstructive pulmonary disease (COPD) caused by air pollution, and develop the corresponding mobile medical assistant system. Through the cross fusion of existing information technology and medical research results, an auxiliary medical system is formed for information recording, tracking tools, early warning model and clinical diagnosis of patients with COPD.

DETAILED DESCRIPTION:
Objective to establish a real-time early warning model of acute exacerbation of chronic obstructive pulmonary disease (COPD) caused by air pollution, and develop the corresponding mobile medical assistant system. Through the cross fusion of existing information technology and medical research results, an auxiliary medical system is formed for information recording, tracking tools, early warning model and clinical diagnosis of patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 40 and < 80 years with post-bronchodilator FEV1/ forced vital capacity (FVC) < 0.7 and percentage predicted of FEV1>30%, who were no exacerbation of symptoms in the 6 weeks preceding the study, were included in the study.

Exclusion Criteria:

* Patients who were diagnosed with other chronic respiratory diseases, including bronchial asthma, bronchiectasis and lung abscess.
* Patients with near-terminal illness, congestive heart failure (NYHA III-IV), or cannot record CAT score timely were excluded.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stable chronic obstructive pulmonary disease (COPD) patients
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-23 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Frequency of acute exacerbations | 1 year incidence rate
  Frequency of acute exacerbations

CONTACTS AND LOCATIONS:
Overall Officials: Yahong Chen, Dr., Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No